CLINICAL TRIAL: NCT02996487
Title: Screening to Prophylax Against Clostridium Difficile Infection
Brief Title: Screening to Prophylax Against Clostridium Difficile Infection -
Acronym: StoP CDI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Matthew Sims, MD, PhD, Director Infectious Disease Research, Beaumont Health; Professor of Internal Medicine and Foundational Medical Studies, OUWB School of Medicine, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2016-254
Record Dates: First submitted 2016-11-17; First posted 2016-12-19 (Estimated); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo every 6 hours. A placebo will look like the drug being studied, but have no active ingredients, in this case it will be fruit punch with vitamins added to mimic the taste of vancomycin.
  Interventions: Other: Placebo
- vancomycin (Active Comparator): Vancomycin 125 mg by mouth every 6 hours
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin
  Arms: vancomycin
Other: Placebo
  Arms: Placebo

SUMMARY:
The goal of this study is to evaluate whether using vancomycin orally can prevent CDI in patients who are colonized with C. difficile who are admitted to the hospital and need antibiotics for another infection.

DETAILED DESCRIPTION:
Screening to Prophylax against CDI (SToP CDI) is a prospective, single-center, double-blinded, randomized, placebo-controlled study of the effectiveness of vancomycin vs. placebo for preventing CDI in patients colonized with toxigenic C. difficile and receiving high-risk antibiotics. The investigators plan to screen 2500 patients to randomize 200.

Consented patients will have a stool sample collected and tested for presence of toxigenic C. difficile by polymerase chain reaction (PCR) test. Patients who test negative will simply be followed for development, severity and outcome of CDI. Patients who test positive (are colonized with C. difficile) will be randomized to one of two arms:

Arm 1: Patients receive 125 mg vancomycin by mouth (PO) every 6 hours as prophylaxis against C. difficile for the duration of their antibiotic treatment +3 days.

Arm 2: Patients receive placebo by mouth (PO) every 6 hours for the duration of their antibiotic treatment +3 days.

ELIGIBILITY:
Inclusion Criteria:

1. Expected duration of admission sufficient to complete screening and enrollment
2. Age ≥18
3. Able to give informed consent
4. Initiated on one of the following antibiotics within the prior 72 hours with an expected duration of at least 72 hours from enrollment: clindamycin, ampicillin, ampicillin/sulbactam, amoxicillin, amoxicillin/clavulanate, moxifloxacin, levofloxacin, piperacillin/tazobactam, or any cephalosporin
5. Maximum expected duration of antibiotics 8 weeks
6. Able to take oral study medications
7. Able to provide a stool sample during hospitalization or within 3 days of discharge
8. Reasonably expected to be able to complete follow up

Exclusion Criteria:

1. Chron's disease, ulcerative colitis, celiac disease, or other chronic diarrheal illness
2. CDI within prior 90 days
3. Currently on metronidazole, oral vancomycin, rifaximin, fidaxomicin, or any other antibiotic active against C. difficile
4. Current diarrhea
5. Current ileostomy, colostomy or other form of surgically disconnected gut such that oral therapy would not be expected to reach the entire lumen of the gut
6. Pregnancy or breast feeding (determined prior to randomization)
7. Travel to an area of endemic diarrheal illness within the last 30 days
8. Life expectancy of less than 60 days
9. Known allergy to vancomycin
10. Participation with other research trials that could impact the results of this trial within the last 30 days
11. Previously enrolled in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1294 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Sims, MD PhD, Principal Investigator — Beaumont Health
Locations (3):
- United States (3):
  - William Beaumont Hospital, Dearborn, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital, Troy, Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on initiation of high-risk antibiotic treatment for a minimum expedited duration of three days, between December 15, 2016 and June 30, 2023. The first participant was enrolled on December 19, 2016 and the last participant was enrolled June 28, 2023.
Pre-assignment Details: Of 1294 participants consented, 728 provided stool samples. 81 met inclusion criteria of culture of stool sample verifying presence of toxigenic C. difficile, and of these 81, 27 consented to randomization to treatment with vancomycin or placebo. These 27 participants are listed in the randomized participant flow below (placebo group or vancomycin group). 647 participants who screened negative and who were not randomized were available for analysis for secondary outcome 5.
Groups:
- Placebo: Patients who screened positive for the presence of C. difficile colonization were randomized to one of two groups: The Placebo group received a placebo liquid every 6 hours. A placebo will look like the drug being studied, but have no active ingredients, in this case it will be fruit punch with vitamins added to mimic the taste of vancomycin.
  Placebo
- Vancomycin: Patients who screened positive for the presence of C. difficile colonization were randomized to one of two groups: the Study group received Vancomycin 125 mg by mouth every 6 hours
  Vancomycin
- Screened Negative for C. Difficile Colonization: Patients who screened negative at enrollment for the presence of C. difficile were not eligible for the randomized portion of the trial, but were available analysis of secondary outcome 5.
Period: Overall Study
Arm/Group | Placebo | Vancomycin | Screened Negative for C. Difficile Colonization
Started | 14 | 13 | 647
Completed | 11 | 8 | 647
Not Completed | 3 | 5 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vancomycin | Screened Negative for C. Difficile Colonization | Total
Number analyzed (Participants) | 14 | 13 | 647 | 674
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 647 patients who screened negative for C. difficile infection and were not enrolled in the randomized portion of the study did not have any baseline characteristics collected except region of enrollment.
  years
    number analyzed (Participants) | 14 | 13 | 0 | 27
    (all) | 63.8 (15.3) | 68.6 (15.5) |  | 68.44 (17.57)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 647 patients who screened negative for C. difficile infection and were not enrolled in the randomized portion of the study did not have any baseline characteristics collected except region of enrollment.
  Participants
    number analyzed (Participants) | 14 | 13 | 0 | 27
    Female | 8 | 6 |  | 14
    Male | 6 | 7 |  | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 647 patients who screened negative for C. difficile infection and were not enrolled in the randomized portion of the study did not have any baseline characteristics collected except region of enrollment.
  Participants
    number analyzed (Participants) | 14 | 13 | 0 | 27
    Hispanic or Latino | 0 | 0 |  | 0
    Not Hispanic or Latino | 12 | 13 |  | 25
    Unknown or Not Reported | 2 | 0 |  | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 647 patients who screened negative for C. difficile infection and were not enrolled in the randomized portion of the study did not have any baseline characteristics collected except region of enrollment.
  Participants
    number analyzed (Participants) | 14 | 13 | 0 | 27
    American Indian or Alaska Native | 0 | 0 |  | 0
    Asian | 0 | 0 |  | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
    Black or African American | 0 | 1 |  | 1
    White | 13 | 12 |  | 25
    More than one race | 0 | 0 |  | 0
    Unknown or Not Reported | 1 | 0 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 647 | 27

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of CDI in Inpatients Receiving Vancomycin Prophylaxis vs. Placebo Who Are on High-risk Antibiotics and Are Colonized With Toxigenic C. Difficile.
Description: Number of participants with CDI in this subgroup of patients as assessed by clinical presentation, polymerase chain reaction (PCR) testing of stool, and EIA test for production of toxins. Patients are considered to have CDI if they have a positive PCR test, a positive toxin enzyme immunoassay (EIA) test, and clinical symptoms compatible with CDI. This outcome is only applicable to the two randomized arms.
Time Frame: 12 weeks after treatment
Population: Data not available for 3 patients lost to follow-up/withdrawn in placebo arm and 4 patients lost to follow-up/withdrawn and 1 death in vancomycin arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vancomycin
Number analyzed (Participants) | 11 | 8
Participants | 0 | 0

2. Secondary Outcome: The Severity of CDI in Patients Receiving Vancomycin Prophylaxis vs. Placebo.
Description: Number of randomized participants with mild, moderate, severe or fulminant disease after treatment. This outcome is only applicable to the two randomized arms.
Time Frame: 12 weeks after treatment
Population: Data not available for 3 patients withdrawn/lost to follow-up in placebo arm and 4 patients withdrawn/lost to follow-up and 1 death in vancomycin arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vancomycin
Number analyzed (Participants) | 11 | 8
Participants
  mild | 0 | 0
  moderate | 0 | 0
  severe | 0 | 0
  fulminant | 0 | 0
  no disease | 11 | 8

3. Secondary Outcome: The Outcome of CDI in Patients Receiving Vancomycin Prophylaxis vs. Placebo.
Description: Number of participants who developed C difficile infection after treatment. This outcome is only applicable to the two randomized arms.
Time Frame: 12 weeks after treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vancomycin
Number analyzed (Participants) | 11 | 8
Participants | 0 | 0

4. Secondary Outcome: The Prevalence of Toxigenic C. Difficile Colonization Among the Inpatient Population Treated With High-risk Antibiotics Based on C. Difficile PCR.
Description: Number of participants who remained colonized with C. difficile after treatment. This outcome is only applicable to the two randomized arms.
Time Frame: 12 weeks after treatment
Population: Data not available for 3 patients withdrawn/lost to follow-up in the placebo arm, and 4 patients withdrawn/lost to follow-up plus one death in the vancomycin arm. One patient in the placebo arm did not give a stool sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Vancomycin
Number analyzed (Participants) | 10 | 8
Participants | 5 | 5

5. Secondary Outcome: The Incidence of CDI in Patients Initiated on High Risk Antibiotics Who Are Not Colonized With Toxigenic C. Difficile.
Description: Number of participants who developed CDI in this subgroup of patients as assessed by clinical presentation and PCR testing of stool. Patients are considered to have CDI if they have a positive PCR test and clinical symptoms compatible with CDI.
Time Frame: 12 weeks after antibiotics
Population: Patients were originally screened for C. difficile colonization prior to randomization. This population represents the 647 participants who initially screened negative for C. difficile colonization and were not placed into the randomized portion of the study, but were assessed at 12 weeks for C. difficile infection. This outcome is not applicable to the colonized, randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Screened Negative for C. Difficile Colonization
Number analyzed (Participants) | 647
Participants | 4

ADVERSE EVENTS:
Time Frame: 12 weeks following completion of antibiotic treatment (an average of 13 weeks total)
Description: Per protocol, not all adverse events were documented. Participants were queried about any current abdominal pain, nausea, vomiting, abdominal bloating, diarrhea, fever; any signs of adverse reaction to the study medication. Adverse events were queried at follow up visits and by participant self-report if it was between follow-up calls.
  Adverse events were not collected for participants who screened negative for C. difficile infection (non-randomized participants); therefore arm not included.
Arm/Group | Placebo | Vancomycin
All-Cause Mortality (participants affected / at risk) | 0/14 | 1/13
Serious Adverse Events (participants affected / at risk) | 4/14 | 4/13
Other Adverse Events (participants affected / at risk) | 8/14 | 8/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=14) | Vancomycin (N=13)
Acute hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute hypoxemic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyponatremia (present at baseline) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gastrointestinal bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bloody diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=14) | Vancomycin (N=13)
Abdominal pain due to constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bruise, left breast (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fall, related to previous issue with right knee (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Left lower quadrant tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fall, with participant hitting head while anticoagulated (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Phlebitis/cellulitis (Vascular disorders) | 0 (0) | 1 (1)
Purulent drainage of left knee incision (Infections and infestations) | 1 (1) | 0 (0)
Infected tooth, required extraction and antibiotic prescription (Infections and infestations) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT02996487/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT02996487/ICF_000.pdf